CLINICAL TRIAL: NCT03038867
Title: Impact of Duloxetine on Male Fertility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1603017099
Record Dates: First submitted 2017-01-27; First posted 2017-02-01 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Infertility, Male; Depression
MeSH Terms: conditions — Infertility, Male; Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Blinded, placebo-controlled, randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, investigator, and outcomes assessor are all blinded to participant's assigned group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duloxetine (Experimental): Duloxetine orally 60mg daily for 5 weeks, then taper to 30mg daily for 1 week
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Duloxetine orally 60mg daily for 5 weeks, then taper to 30mg daily for 1 week
  Arms: Duloxetine
Drug: Placebo — Placebo orally 2 tabs daily for 5 weeks, then taper to 1 tab daily for 1 week
  Arms: Placebo

SUMMARY:
The investigators are conducting a placebo-controlled, randomized control trial with duloxetine in healthy, fertile men not previously on any antidepressants. Participants will be randomized to either the duloxetine or placebo groups for 6 weeks. The investigators will assess changes in sperm DNA fragmentation at 0, 2, 6, 8, and 10 weeks. Other outcomes measured will include semen parameters (sperm concentration, motility, morphology), hormone levels (testosterone, estrogen, prolactin, LH, FSH), and sexual function (IIEF and MSHQ) surveys.

DETAILED DESCRIPTION:
Antidepressant medications are commonly prescribed in the USA not only for depression, but also for anxiety disorders such as generalized anxiety disorder and obsessive-compulsive disorder, premature ejaculation, post-traumatic stress disorder, and neuropathic pain. Despite being widely prescribed in the United States in men of reproductive age, the impact of antidepressants on fertility has not been extensively studied.

After noticing worsened semen parameters in men on anti-depressants, the investigators performed the first prospective study to demonstrate a deleterious impact of selective serotonin reuptake inhibitors (SSRI) on sperm DNA integrity, which has been linked to reproductive outcomes. Further small studies have corroborated the negative impact of SSRIs on male fertility, as assessed by semen parameters and/or sperm DNA integrity.

No studies have examined the impact of a newer, but similar, class of antidepressant - the serotonin-norepinephrine reuptake inhibitor (SNRI). Like SSRIs, SNRIs inhibit the reuptake of serotonin, but also act on norepinephrine. The use of SNRIs has increased recently due to their slightly improved efficacy profile when compared to SSRIs. Duloxetine is an SNRI and is one of the most commonly prescribed anti-depressants in the United States.

The investigators are conducting this trial to determine whether or not the administration of duloxetine will result in a deterioration in sperm DNA fragmentation in healthy, fertile men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged 18-65 years old;
* normal or borderline semen analysis (sperm concentration > 10 million/mL, sperm motility > 30%, sperm morphology > 3%);
* willing to engage in sexual activity (alone or with a partner) at least once per week for the duration of the study;
* capable of providing semen sample.

Exclusion Criteria:

* Clinically detected varicocele;
* oligoasthenoteratospermia or azoospermia on semen analysis;
* ongoing attempts to initiate pregnancy;
* current sexual dysfunction (classified as moderate or worse on IIEF);
* history of seizure disorder;
* history of previous chemotherapy or radiation therapy;
* current psychiatric history or history of bipolar disorder;
* family history of bipolar disorder, depression, or suicide;
* use of any psychotropic medications or anticonvulsants;
* use of sleeping pills more than once per week;
* use of any hormonal medications on a daily or intermittent basis during the preceding 3 months;
* use of medications which may affect hormone measures and/or sexual function;
* inability to read, follow instructions, or complete questionnaires in English;
* consumption of tobacco or illicit drugs;
* consumption of >2oz of alcohol daily.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schlegel, MD, Study Chair — Weill Medical College of Cornell University; Nahid Punjani, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 37 | 32
Completed | 37 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 37 | 32 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 32 | 69
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 37 | 32 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 32 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abnormal Sperm DNA Fragmentation at 6 Weeks
Description: Number of participants with TUNEL values > 25% at 6 weeks in each treatment group
Time Frame: 6 Weeks (primary time point of interest)
Population: 11 patients in the Duloxetine group and 7 patients in the Placebo group did not have Tunel data measured at 6 weeks (patients were not available).
Measure: Count of Participants; unit: Participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 25
Participants | 0 | 2

2. Primary Outcome: Number of Participants With Abnormal Sperm DNA Fragmentation at 0 Weeks
Description: Number of participants with Tunel Values > 25% at 0 Weeks (baseline) in each treatment group
Time Frame: 0 weeks
Population: 5 patients in the Duloxetine group did not have Tunel data measured at 0 weeks (patients were not available)
Measure: Count of Participants; unit: Participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 32 | 32
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Sperm DNA Fragmentation at 2 Weeks
Description: Number of participants with Tunel values > 25% at 2 weeks in each treatment group
Time Frame: 2 weeks
Population: 12 patients in the Duloxetine group and 2 patients in the Placebo group did not have Tunel data at 2 weeks (patients were not available).
Measure: Count of Participants; unit: Participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 25 | 30
Participants | 1 | 2

4. Primary Outcome: Number of Participants With Abnormal Sperm DNA Fragmentation at 8 Weeks
Description: Number of participants with Tunel values > 25% at 8 weeks in each treatment group
Time Frame: 8 weeks
Population: 15 patients in the Duloxetine group and 4 patients in the Placebo group did not have Tunel data at 8 weeks (patients were not available).
Measure: Count of Participants; unit: Participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 22 | 28
Participants | 1 | 0

5. Primary Outcome: Number of Participants With Abnormal Sperm DNA Fragmentation at 10 Weeks
Description: Number of participants with Tunel values > 25% at 10 weeks in each treatment group
Time Frame: 10 Weeks
Population: 18 patients in the Duloxetine group and 4 patients in the Placebo group did not have Tunel data at 10 weeks (patients were not available).
Measure: Count of Participants; unit: Participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 19 | 28
Participants | 0 | 2

6. Secondary Outcome: Sperm Concentration at 0 Weeks
Description: Sperm concentration (number of sperm/mL) in semen analysis at 0 weeks
Time Frame: 0 weeks
Population: 3 patients in the Duloxetine group did not have sperm concentration measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: Number of sperm/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 34 | 32
Number of sperm/mL | 57.4 (40.3) | 50.2 (33.4)

7. Secondary Outcome: Sperm Concentration at 2 Weeks
Description: Sperm concentration (number of sperm/mL) in semen analysis at 2 weeks
Time Frame: 2 weeks
Population: 10 patients in the Duloxetine group and 2 patients in the Placebo group did not have sperm concentration measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: Number of sperm/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 27 | 30
Number of sperm/mL | 48.9 (38.7) | 50.0 (41.4)

8. Secondary Outcome: Sperm Concentration at 6 Weeks
Description: Sperm concentration (number of sperm/mL) in semen analysis at 6 weeks
Time Frame: 6 weeks
Population: 11 patients in the Duloxetine group and 5 patients in the Placebo group did not have sperm concentration measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: Number of sperm/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 27
Number of sperm/mL | 44.6 (24.2) | 43.9 (32.5)

9. Secondary Outcome: Sperm Concentration at 8 Weeks
Description: Sperm concentration (number of sperm/mL) in semen analysis at 8 weeks
Time Frame: 8 weeks
Population: 14 patients in the Duloxetine group and 2 patients in the Placebo group did not have sperm concentration measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: Number of sperm/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 23 | 30
Number of sperm/mL | 45.7 (29.8) | 47.1 (28.7)

10. Secondary Outcome: Sperm Concentration at 10 Weeks
Description: Sperm concentration (number of sperm/mL) in semen analysis at 10 weeks
Time Frame: 10 Weeks
Population: 16 patients in the Duloxetine group and 2 patients in the Placebo group did not have sperm concentration measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: Number of sperm/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 21 | 30
Number of sperm/mL | 42.0 (26.3) | 42.7 (26.0)

11. Secondary Outcome: Sperm Motility at 0 Weeks
Description: Sperm motility (mean percent) at 0 weeks
Time Frame: 0 weeks
Population: 3 patients in the Duloxetine group did not have motility measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: percent motility
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 34 | 32
percent motility | 61.7 (9.5) | 59.7 (11.4)

12. Secondary Outcome: Sperm Motility at 2 Weeks
Description: Sperm motility (mean percent) at 2 weeks
Time Frame: 2 weeks
Population: 11 patients in the Duloxetine group and 2 patients in the Placebo group did not have motility measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: percent motility
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 30
percent motility | 54.3 (13.3) | 55.2 (13.4)

13. Secondary Outcome: Sperm Motility at 6 Weeks
Description: Sperm motility (mean percent) at 6 weeks
Time Frame: 6 weeks
Population: 11 patients in the Duloxetine group and 5 patients in the Placebo group did not have motility measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: percent motility
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 27
percent motility | 57.2 (11.2) | 50.4 (20.6)

14. Secondary Outcome: Sperm Motility at 8 Weeks
Description: Sperm motility (mean percent) at 8 weeks
Time Frame: 8 weeks
Population: 13 patients in the Duloxetine group and 2 patients in the Placebo group did not have motility measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: percent motility
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 24 | 30
percent motility | 51.1 (18.6) | 58.5 (12.1)

15. Secondary Outcome: Sperm Motility at 10 Weeks
Description: Sperm motility (mean percent) at 10 weeks
Time Frame: 10 Weeks
Population: 15 patients in the Duloxetine group and 3 patients in the Placebo group did not have motility measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: percent motility
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 22 | 29
percent motility | 54.4 (17.4) | 53.9 (19.7)

16. Secondary Outcome: Sperm Head Defects at 0 Weeks
Description: Sperm head defects (mean number) at 0 weeks
Time Frame: 0 weeks
Population: 3 patients in the Duloxetine group did not have head defects measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 34 | 32
defects | 88.4 (16.0) | 89.9 (8.11)

17. Secondary Outcome: Sperm Head Defects at 2 Weeks
Description: Sperm head defects (mean number) at 2 weeks
Time Frame: 2 weeks
Population: 11 patients in the Duloxetine group and 2 patients in the Placebo group did not have head defects measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 30
defects | 91.5 (4.02) | 90.7 (7.86)

18. Secondary Outcome: Sperm Head Defects at 6 Weeks
Description: Sperm head defects (mean number) at 6 weeks
Time Frame: 6 weeks
Population: 11 patients in the Duloxetine group and 5 patients in the Placebo group did not have head defects measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 27
defects | 91.6 (4.38) | 91.3 (10.1)

19. Secondary Outcome: Sperm Head Defects at 8 Weeks
Description: Sperm head defects (mean number) at 8 weeks
Time Frame: 8 weeks
Population: 13 patients in the Duloxetine group and 2 patients in the Placebo group did not have head defects measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 24 | 30
defects | 92.3 (4.54) | 88.7 (15.1)

20. Secondary Outcome: Sperm Head Defects at 10 Weeks
Description: Sperm head defects (mean number) at 10 weeks
Time Frame: 10 Weeks
Population: 15 patients in the Duloxetine group and 3 patients in the Placebo group did not have head defects measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 22 | 29
defects | 90.8 (5.65) | 88.3 (16.6)

21. Secondary Outcome: Sperm Neck Defects at 0 Weeks
Description: Sperm neck defects (mean number) at 0 weeks
Time Frame: 0 weeks
Population: 3 patients in the Duloxetine group did not have neck defects measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 33 | 32
defects | 1.36 (2.97) | 2.55 (4.47)

22. Secondary Outcome: Sperm Neck Defects at 2 Weeks
Description: Sperm neck defects (mean number) at 2 weeks
Time Frame: 2 weeks
Population: 11 patients in the Duloxetine group and 2 patients in the Placebo group did not have neck defects measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 30
defects | 2.65 (5.83) | 1.00 (3.04)

23. Secondary Outcome: Sperm Neck Defects at 6 Weeks
Description: Sperm neck defects (mean number) at 6 weeks
Time Frame: 6 weeks
Population: 11 patients in the Duloxetine group and 11 patients in the Placebo group did not have neck defects measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 26
defects | 1.12 (4.35) | 0.62 (1.96)

24. Secondary Outcome: Sperm Neck Defects at 8 Weeks
Description: Sperm neck defects (mean number) at 8 weeks
Time Frame: 8 weeks
Population: 14 patients in the Duloxetine group and 2 patients in the Placebo group did not have neck defects measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 23 | 30
defects | 1.17 (2.66) | 0.50 (1.61)

25. Secondary Outcome: Sperm Neck Defects at 10 Weeks
Description: Sperm neck defects (mean number) at 10 weeks
Time Frame: 10 Weeks
Population: 15 patients in the Duloxetine group and 3 patients in the Placebo group did not have neck defects measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 22 | 29
defects | 0.91 (2.72) | 1.55 (3.93)

26. Secondary Outcome: Sperm Tail Defects at 0 Weeks
Description: Sperm tail defects (mean number) at 0 weeks
Time Frame: 0 weeks
Population: 6 patients in the Duloxetine group and 4 patients in the Placebo group did not have tail defects measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 31 | 28
defects | 0.13 (0.72) | 1.89 (7.86)

27. Secondary Outcome: Sperm Tail Defects at 2 Weeks
Description: Sperm tail defects (mean number) at 2 weeks
Time Frame: 2 weeks
Population: 16 patients in the Duloxetine group and 3 patients in the Placebo group did not have tail defects measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 21 | 29
defects | 0.00 (0.00) | 1.66 (7.52)

28. Secondary Outcome: Sperm Tail Defects at 6 Weeks
Description: Sperm tail defects (mean number) at 6 weeks
Time Frame: 6 weeks
Population: 11 patients in the Duloxetine group and 7 patients in the Placebo group did not have tail defects measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 25
defects | 0.04 (0.20) | 2.64 (11.0)

29. Secondary Outcome: Sperm Tail Defects at 8 Weeks
Description: Sperm tail defects (mean number) at 8 weeks
Time Frame: 8 weeks
Population: 14 patients in the Duloxetine group and 4 patients in the Placebo group did not have tail defects measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 23 | 28
defects | 0.35 (1.30) | 1.25 (3.74)

30. Secondary Outcome: Sperm Tail Defects at 10 Weeks
Description: Sperm tail defects (mean number) at 10 weeks
Time Frame: 10 Weeks
Population: 15 patients in the Duloxetine group and 4 patients in the Placebo group did not have tail defects measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: defects
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 22 | 28
defects | 1.09 (5.12) | 0.96 (3.67)

31. Secondary Outcome: Testosterone Level at 0 Weeks
Description: Testosterone level (ng/dL) at 0 weeks
Time Frame: 0 weeks
Population: 3 patients in the Duloxetine group did not have testosterone measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 34 | 32
ng/dL | 464 (165) | 448 (160)

32. Secondary Outcome: Testosterone Level at 2 Weeks
Description: Testosterone level (ng/dL) at 2 weeks
Time Frame: 2 weeks
Population: 8 patients in the Duloxetine group did not have testosterone measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 29 | 32
ng/dL | 431 (126) | 482 (171)

33. Secondary Outcome: Testosterone Level at 6 Weeks
Description: Testosterone level (ng/dL) at 6 weeks
Time Frame: 6 weeks
Population: 12 patients in the Duloxetine group and 2 patients in the Placebo group did not have testosterone measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 25 | 30
ng/dL | 485 (170) | 438 (174)

34. Secondary Outcome: Testosterone Level at 8 Weeks
Description: Testosterone level (ng/dL) at 8 weeks
Time Frame: 8 weeks
Population: 12 patients in the Duloxetine group and 4 patients in the Placebo group did not have testosterone measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 25 | 28
ng/dL | 534 (237) | 460 (144)

35. Secondary Outcome: Testosterone Level at 10 Weeks
Description: Testosterone level (ng/dL) at 10 weeks
Time Frame: 10 Weeks
Population: 21 patients in the Duloxetine group and 8 patients in the Placebo group did not have testosterone measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 16 | 24
ng/dL | 445 (165) | 509 (167)

36. Secondary Outcome: Estrogen Level at 0 Weeks
Description: Estrogen level (pg/mL) at 0 weeks
Time Frame: 0 weeks
Population: 6 patients in the Duloxetine group and 3 patients in the Placebo group did not have estrogen measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 31 | 29
pg/mL | 51.8 (39.4) | 58.5 (51.9)

37. Secondary Outcome: Estrogen Level at 2 Weeks
Description: Estrogen level (pg/mL) at 2 weeks
Time Frame: 2 weeks
Population: 16 patients in the Duloxetine group did not have estrogen measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 25 | 32
pg/mL | 53.0 (37.6) | 44.4 (25.7)

38. Secondary Outcome: Estrogen Level at 6 Weeks
Description: Estrogen level (pg/mL) at 6 weeks
Time Frame: 6 weeks
Population: 16 patients in the Duloxetine group and 5 patients in the Placebo group did not have estrogen measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 21 | 27
pg/mL | 45.8 (30.7) | 43.5 (28.2)

39. Secondary Outcome: Estrogen Level at 8 Weeks
Description: Estrogen level (pg/mL) at 8 weeks
Time Frame: 8 weeks
Population: 17 patients in the Duloxetine group and 6 patients in the Placebo group did not have testosterone measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 20 | 26
pg/mL | 49.3 (31.9) | 39.0 (24.8)

40. Secondary Outcome: Estrogen Level at 10 Weeks
Description: Estrogen level (pg/mL) at 10 weeks
Time Frame: 10 Weeks
Population: 23 patients in the Duloxetine group and 8 patients in the Placebo group did not have estrogen measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 14 | 24
pg/mL | 31.7 (12.2) | 133 (467)

41. Secondary Outcome: Prolactin Level at 0 Weeks
Description: Prolactin level (ng/mL) at 0 weeks
Time Frame: 0 weeks
Population: 3 patients in the Duloxetine group did not have prolactin measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 34 | 32
ng/mL | 11.9 (5.78) | 12.4 (4.85)

42. Secondary Outcome: Prolactin Level at 2 Weeks
Description: Prolactin level (ng/mL) at 2 weeks
Time Frame: 2 weeks
Population: 8 patients in the Duloxetine group did not have prolactin measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 29 | 32
ng/dL | 9.74 (3.69) | 11.3 (6.01)

43. Secondary Outcome: Prolactin Level at 6 Weeks
Description: Prolactin level (ng/mL) at 6 weeks
Time Frame: 6 weeks
Population: 11 patients in the Duloxetine group and 1 patient in the Placebo group did not have prolactin measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 31
ng/mL | 10.3 (5.05) | 9.60 (6.01)

44. Secondary Outcome: Prolactin Level at 8 Weeks
Description: Prolactin level (ng/mL) at 8 weeks
Time Frame: 8 weeks
Population: 12 patients in the Duloxetine group and 2 patients in the Placebo group did not have prolactin measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 25 | 30
ng/mL | 10.1 (4.91) | 8.98 (3.66)

45. Secondary Outcome: Prolactin Level at 10 Weeks
Description: Prolactin level (ng/mL) at 10 weeks
Time Frame: 10 Weeks
Population: 20 patients in the Duloxetine group and 5 patients in the Placebo group did not have prolactin measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 17 | 27
ng/mL | 8.83 (3.31) | 11.6 (6.14)

46. Secondary Outcome: Luteinizing Hormone Level at 0 Weeks
Description: Luteinizing hormone level (mIU/mL) at 0 weeks
Time Frame: 0 weeks
Population: 3 patients in the Duloxetine group did not have LH measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 34 | 32
mIU/mL | 4.11 (4.98) | 3.37 (1.72)

47. Secondary Outcome: Luteinizing Hormone Level at 2 Weeks
Description: Luteinizing hormone level (mIU/mL) at 2 weeks
Time Frame: 2 weeks
Population: 8 patients in the Duloxetine group did not have LH measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 29 | 32
mIU/mL | 4.00 (5.47) | 3.57 (1.55)

48. Secondary Outcome: Luteinizing Hormone Level at 6 Weeks
Description: Luteinizing hormone level (mIU/mL) at 6 weeks
Time Frame: 6 weeks
Population: 11 patients in the Duloxetine group and 1 patient in the Placebo group did not have LH measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 26 | 31
mIU/mL | 4.51 (5.92) | 3.42 (1.43)

49. Secondary Outcome: Luteinizing Hormone Level at 8 Weeks
Description: Luteinizing hormone level (mIU/mL) at 8 weeks
Time Frame: 8 weeks
Population: 13 patients in the Duloxetine group and 2 patients in the Placebo group did not have LH measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 24 | 30
mIU/mL | 4.18 (5.50) | 3.70 (1.42)

50. Secondary Outcome: Luteinizing Hormone Level at 10 Weeks
Description: Luteinizing hormone level (mIU/mL) at 10 weeks
Time Frame: 10 Weeks
Population: 22 patients in the Duloxetine group and 5 patients in the Placebo group did not have LH measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 15 | 27
mIU/mL | 4.98 (6.40) | 3.78 (1.48)

51. Secondary Outcome: Follicle Stimulating Hormone Level at 0 Weeks
Description: Follicle stimulating hormone level (mIU/mL) at 0 weeks
Time Frame: 0 weeks
Population: 5 patients in the Duloxetine group and 1 patient in the Placebo group did not have FSH measured at 0 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 32 | 31
mIU/mL | 6.56 (12.3) | 5.26 (4.30)

52. Secondary Outcome: Follicle Stimulating Hormone Level at 2 Weeks
Description: Follicle stimulating hormone level (mIU/mL) at 2 weeks
Time Frame: 2 weeks
Population: 9 patients in the Duloxetine group and 1 patient in the Placebo group did not have FSH measured at 2 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 28 | 31
mIU/mL | 5.56 (5.86) | 5.30 (4.27)

53. Secondary Outcome: Follicle Stimulating Hormone Level at 6 Weeks
Description: Follicle stimulating hormone level (mIU/mL) at 6 weeks
Time Frame: 6 weeks
Population: 16 patients in the Duloxetine group and 2 patients in the Placebo group did not have FSH measured at 6 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 21 | 30
mIU/mL | 4.57 (5.71) | 5.14 (4.39)

54. Secondary Outcome: Follicle Stimulating Hormone Level at 8 Weeks
Description: Follicle stimulating hormone level (mIU/mL) at 8 weeks
Time Frame: 8 weeks
Population: 15 patients in the Duloxetine group and 4 patients in the Placebo group did not have FSH measured at 8 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 22 | 28
mIU/mL | 4.18 (3.97) | 5.29 (3.71)

55. Secondary Outcome: Follicle Stimulating Hormone Level at 10 Weeks
Description: Follicle stimulating hormone level (mIU/mL) at 10 weeks
Time Frame: 10 Weeks
Population: 23 patients in the Duloxetine group and 6 patients in the Placebo group did not have FSH measured at 10 weeks (patients were not available).
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 14 | 26
mIU/mL | 5.54 (5.44) | 5.95 (5.43)

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Arm/Group | Duloxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/32
Other Adverse Events (participants affected / at risk) | 0/37 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT03038867/Prot_SAP_000.pdf